CLINICAL TRIAL: NCT04756180
Title: A Placebo-Controlled, Multicenter, Randomized, Double-Blind, Parallel Group Study to Investigate the Efficacy and Safety of Omega-3-acid Ethyl Ester Over 12 Weeks in Chinese Subjects With Hypertriglyceridemia
Brief Title: An Efficacy and Safety Study of Omega-3-acid Ethyl Ester in Chinese Subjects With Hypertriglyceridemia.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUFA3001
Record Dates: First submitted 2021-01-12; First posted 2021-02-16 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Hypertriglyceridemia
MeSH Terms: conditions — Hypertriglyceridemia

STUDY DESIGN:
Masking Description: Double Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omacor (Experimental): Omacor 2gm/day for first 4 week followed by 4gms/day for 8 weeks
  Interventions: Drug: Omega-3-acid ethyl ester or Placebo
- Placebo (Placebo Comparator): Omacor Placebo 2gm/day for first 4 week followed by 4gms/day for 8 weeks
  Interventions: Drug: Omega-3-acid ethyl ester or Placebo

INTERVENTIONS:
Drug: Omega-3-acid ethyl ester or Placebo — Omega-3-acid ethyl ester 2 gm/day for first 4 week followed by 4gm/day for 8 week

SUMMARY:
The primary objective was to investigate the effect of 12-week treatment of Omacor on fasting serum triglycerides (TG) in Chinese subjects with hypertriglyceridemia (HTG). The secondary objectives were to investigate the safety and tolerability and effect of Omacor on lipid parameters after 12 weeks treatment.

DETAILED DESCRIPTION:
This was a multicenter, randomized, double-blind, parallel-group study of twice daily treatment of Omacor or matching placebo in subjects with moderate or severe HTG.

ELIGIBILITY:
Inclusion Criteria:

* Baseline fasting serum TG level > 200mg/dL and <1000mg/dL, in subjects treated for HTG.
* If on previous statin therapy, the treatment should have been kept stable in the last 3 months before entering the study.
* Able and willing to give written informed consent.

Exclusion Criteria:

* Subjects taking fish oil capsules 8 weeks prior to inclusion in this study.
* Known allergy to the active ingredient, or fish, soya, corn or olive oild (placebos).
* Pregnant of lactating females.
* Known increased risk of hemorrhage such as recent surgery, gastrointestinal hemorrhagic disease.
* Significant hepatic disease.
* Significantly reduced renal function.
* Alcohol consumption >30g for male and 20g for female daily.
* Concomitant use of other investigational drugs.
* Subject related to the investigator.
* Subject expected to be not compliant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Percent change in fasting serum TG | Baseline to end of treatment at treatment week 12
  Percent change from baseline in fasting serum TG

SECONDARY OUTCOMES:
Change in total cholesterol, LDL-cholesterol, HDL cholesterol, non-HDL-cholesterol and the LDL/HDL ratio | Between baseline and end of treatment week 12
  Change from baseline in total cholesterol, LDL-cholesterol, HDL cholesterol, non-HDL-cholesterol and the LDL/HDL ratio

CONTACTS AND LOCATIONS:
Overall Officials: Pooi Lee Chin, Study Director — Abbott

IPD SHARING:
Plan to Share IPD: No